CLINICAL TRIAL: NCT07129564
Title: Effects on Sinus Rhythm Maintenance and Atrial Remodeling After Cardioversion of Persistent Atrial Fibrillation: a Prospective, Multi-center, Cohort Study-stepwise Strategy for Treatment of Atrialfibrillation Substrate Study
Brief Title: Stepwise Strategy for Treatment of Atrialfibrillation Substrate Study
Acronym: SAFE
Status: Recruiting | Type: Observational
Sponsor: Yuehui Yin (Other)
Responsible Party: Sponsor-Investigator, Yuehui Yin, MD, The Second Affiliated Hospital of Chongqing Medical University
Organization: The Second Affiliated Hospital of Chongqing Medical University (Other)
Other Study IDs: SAFE study
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- reversed: at least a 15% reduction in the max LA volume
  Interventions: Other: treatment react
- non-reversed: less than 15% reduction in the max LA volume

INTERVENTIONS:
Other: treatment react — Reverse remodeling of the LA was defined as at least a 15% reduction in the max LA volume after electrical or pharmacological cardioversion for 3 months
  Groups: reversed

SUMMARY:
Electrical/pharmacological cardioversion improves structural remodeling of left atrium. We hypothesized that radiofrequency ablation surgery for atrial fibrillation has a higher success rate and a lower recurrence rate of atrial fibrillation in patients with improved atrial stroma. This study is a multicenter, prospective, observational study conducted in China to evaluate whether sacubitril/valsartan can reduce atrial fibrillation recurrence rates, improve cardiac structure and function, and analyze the factors influencing the maintenance rate of sinus rhythm after atrial fibrillation ablation.

DETAILED DESCRIPTION:
Background: Atrial fibrillation (AF) is associated with significant co-morbidities such as embolic stroke, heart failure, dementia. Consequently, AF poses a significant burden to the healthcare system, in both direct and indirect costs. The management of AF is complex, especially for patients with persistent AF. It is preferable to terminate the AF and restore normal sinus rhythm for relief of symptoms associated with AF or improvement of cardiac structure and function. The maintenance of AF, especially persist AF is associated with fibrosis of left atria. Furthermore, AF itself promotes fibrosis, which in turn leads to increased conduction heterogeneity within the atrial substrate resulting in further progression of AF. In animal models, alterations in myocytes after sustained AF resemble those of myocardial hibernation. Ultimately, these structural changes would lead to Calcium overload and metabolic stress, similar changes have been observed in humans. In humans, atrial dilatation and degenerative changes have been observed. Interstitial fibrosis is the prime cause of structural remodeling in left atrium. Whether reversal of sinus rhythm can reverse fibrosis partly? The introduction of Late Gadolinium enhancement magnetic resonance imaging (LGE-MRI) sequence now allows for non-invasive and dynamic assessment of the location and extent of atrial fibrosis.

The investigators propose to evaluate whether sacubitril/valsartan can reduce atrial fibrillation recurrence rates, improve cardiac structure and function, and analyze the factors influencing the maintenance rate of sinus rhythm after atrial fibrillation ablation.

Objectives:

Primary: In patients with persistent atrial fibrillation and left atrial enlargement, the first part: after drug or electrical cardioversion, on the basis of using amiodarone to maintain sinus rhythm, they were divided into the group prescribed sacubitril/valsartan and the control group, and evaluated whether sacubitril/valsartan could reduce the recurrence rate of atrial fibrillation, improve cardiac structure and function, and improve atrial fibrosis by comparing the maintenance rate of sinus rhythm after cardioversion, ultrasound assessment of atrial structure and function, cardiac MRI evaluation of cardiac structure, function and fibrosis.

The second part: Combined with the patient's wishes, researchers perform annular pulmonary vein isolation 3 to 6 months after cardioversion, evaluate the patient's sinus rhythm maintenance rate and cardiac structure and function at 3 months, 6 months, 1 year and 2 years after ablation. Then we will evaluate whether the improvement of atrial structure and function before surgery can predict the success rate of surgery, and evaluate whether sacubitril/valsartan further improves the success rate of surgery compared with the control group. If the number of patients in the subgroup is sufficient, subgroup analysis can be performed in a specific patient subgroup。

Secondary:

We will assess the effects on patients with the following outcomes, including: analysis of other factors influencing left atrial remodeling. The influencing factors will be analyze of sinus rhythm maintenance rate after other electrical cardioversion.If the number of patients in the subgroup is sufficient, subgroup analysis can be performed in a specific subgroup of patients

ELIGIBILITY:
Inclusion Criteria:

Aged 18-80 years, with persistent atrial fibrillation complicated by left atrial enlargement (left atrial anteroposterior diameter 40-50mm); Having the willingness to undergo atrial fibrillation cardioversion and planned to receive amiodarone for pharmacological cardioversion; Having signed a written informed consent form for participation in the study; Not concurrently participating in any other interventional studies.

Exclusion Criteria:

Females who are pregnant, lactating, or planning to have children within the next 2 years; Patients whose arrhythmia fails to convert to sinus rhythm with medication and who refuse electrical cardioversion; Patients whose arrhythmia cannot be converted to sinus rhythm with either medication or electrical cardioversion; Glomerular filtration rate (eGFR) < 30 ml/min/1.73m² (calculated by the CKD-EPI formula); Patients with biliary cirrhosis or cholestasis; Hyperthyroidism; A history of bradycardia (heart rate < 50 beats/min) or atrioventricular block of second degree or higher; Sick sinus syndrome; Known allergy to iodine, amiodarone, or any of its excipients; Concomitant use of other drugs that prolong the QT interval, or a history of torsades de pointes; Contraindications to atrial fibrillation cardioversion, such as cardiac thrombosis or contraindications to anticoagulation;

A history or current presence of the following diseases or conditions:

1. Moderate to severe rheumatic heart disease, valvular heart disease; a history of atrial-related surgery, including valve replacement, radiofrequency ablation for atrial fibrillation/atrial tachycardia/atrial flutter, atrial septal defect occlusion, or complex congenital heart disease surgery;
2. A history of myocardial infarction, unstable angina, syncope, or cerebrovascular accident within 3 months;
3. NYHA Class III-IV congestive heart failure or EF < 40%;
4. Patients judged by the investigator to have poor compliance, inability to complete the study as required, or an expected lifespan of less than 1 year.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: persistent atrial fibrillation with left atrial enlargement
Sampling Method: Non-Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2023-04-27 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
recurrence of atrial tachyarrhythmia | 1 year
  the first documented recurrence of any atrial tachyarrhythmia (atrial fibrillation, atrial flutter, or atrial tachycardia) between 91 and 365 days after catheter ablation or the initiation of an antiarrhythmic drug

CONTACTS AND LOCATIONS:
Locations (1):
- the second affiliated hospital of CQMU, Chongqing, China

IPD SHARING:
Plan to Share IPD: No
Sharing such data without the patient's explicit authorization may violate their right to privacy and contravene the informed consent terms obtained in the study.